CLINICAL TRIAL: NCT07387393
Title: Peau o le Vasa: Accelerating the Currents of Health Advances for Pasifika People
Brief Title: To Test the Effectiveness and Implementation Approach of a 3-month PILI Pasifika Program Lifestyle Program With Components of Social Determinants of Health Activities in Real-world Settings (Clinical and Non-clinical Settings) Across 3 Years
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Association of Pasifika Organizations (Unknown); Papa Ola Lōkahi (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Peau o le Vasa Phase II; OT2HL158287 (NIH)
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Cardiometabolic Conditions; Hypertension (HTN); Dyslipidemia; Pre-diabetes; Type 2 Diabetes Mellitus (T2DM); Overweight (BMI > 25); Weight Loss Trial
Keywords: Weight Loss Intervention; CHWs; Community Health Workers; PILI Lifestyle Program; Social Determinants of Health; U.S. Pacific Jurisdictions; Continental U.S.; Pacific Islands; Hawai'i; Education; Lifestyle Intervention; Community-Based Participatory Research (CBPR); Academic and Community Partnership; Native Hawaiians; Pacific Islanders; PILI Pasifika Program; PPP
MeSH Terms: conditions — Hypertension; Dyslipidemias; Glucose Intolerance; Diabetes Mellitus, Type 2; Overweight

STUDY DESIGN:
Intervention Model Description: Multisite, cluster-randomized implementation trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PILI Pasifika Program - Standard Facilitation (Active Comparator): Participants in the Standard Facilitation group will engage in a 3-month PILI Pasifika Program (PPP) with a trained Community Health Worker (CHW). Each week during the 3-months, participants will meet for approximately 1-1.5 hours to receive a Weekly Lesson or engage in an SDoH activity. Participants will also complete an assessment at baseline, at the 3-month program completion, and at the 9-month follow-up.
  Interventions: Behavioral: PILI (Partnership for Improving Lifestyle Intervention) Pasifika Program - Standard Facilitation
- PILI Pasifika Program - Enhanced Facilitation (Experimental): Participants in the Enhanced Facilitation group will engage in a 3-month PILI Pasifika Program (PPP) with a trained Community Health Worker (CHW). Each week during the 3-month period, participants will meet for approximately 1-1.5 hours to receive a Weekly Lesson or engage in an SDoH activity. CHWs managing participants in the Enhanced Facilitation group may receive additional support to strengthen program fit, problem-solving, and uptake across diverse settings, offering participants more tailored guidance. Participants will also complete an assessment at baseline, at 3-month program completion, and at the 9-month follow-up.
  Interventions: Behavioral: PILI (Partnership for Improving Lifestyle Intervention) Pasifika Program - Enhanced Facilitation

INTERVENTIONS:
Behavioral: PILI (Partnership for Improving Lifestyle Intervention) Pasifika Program - Standard Facilitation — The PILI Pasifika Program (PPP) is an adapted 3-month behavioral lifestyle intervention with an enhanced social determinants of health (SDOH) component focused on initiating weight loss and addressing social and cultural challenges, such as access to healthy foods, housing, and employment issues, among Native Hawaiians and Pacific Islanders (NHPIs). The 3-month PPP includes 8 lessons that offer empirically supported strategies (e.g., plate method, stimulus control), grounded in Social Cognitive Theory, to improve healthy eating, physical activity, and time and stress management, as well as 4 SDOH activities that provide guidance on community needs such as food access, transportation, and housing throughout the program. Standard Facilitation is to be implemented.
  Other Names: PPP; PILI Pasifika Program; Partnership for Improving Lifestyle Intervention (PILI) + Social Determinants of Health Component; PPP-SF
  Arms: PILI Pasifika Program - Standard Facilitation
Behavioral: PILI (Partnership for Improving Lifestyle Intervention) Pasifika Program - Enhanced Facilitation — The PILI Pasifika Program (PPP) is an adapted 3-month behavioral lifestyle intervention with an enhanced social determinants of health (SDOH) component focused on initiating weight loss and addressing social and cultural challenges, such as access to healthy foods, housing, and employment issues, among Native Hawaiians and Pacific Islanders (NHPIs). The 3-month PPP includes 8 lessons that offer empirically supported strategies (e.g., plate method, stimulus control), grounded in Social Cognitive Theory, to improve healthy eating, physical activity, and time and stress management, as well as 4 SDOH activities that provide guidance on community needs such as food access, transportation, and housing throughout the program. In this enhanced facilitation intervention, we are utilizing a peer coach CHW to provide additional support to CHWs to strengthen program fit, problem-solving, and uptake across diverse settings, offering participants more tailored guidance.
  Other Names: Partnership for Improving Lifestyle Intervention (PILI) + Social Determinants of Health Component; PPP; PILI Pasifika Program; PPP-EF
  Arms: PILI Pasifika Program - Enhanced Facilitation

SUMMARY:
In this study, the investigators are testing the effectiveness and implementation of the Community Health Workers (CHW)-delivered PILI Pasifika Program (PPP) Standard Facilitation or Enhanced Facilitation across 3 regions, the U.S. Affiliated Pacific Islands (USAPI), the continental U.S., and Hawai'i, among 600 Native Hawaiian and Pacific Islander (NHPI) participants in two settings, (clinical and non-clinical) over a 3-year period. The PPP is a 3-month lifestyle intervention that includes a Social Determinants of Health (SDOH) component and was NHPI-adapted from the Diabetes Prevention Program's Lifestyle Program, renamed to the PILI Lifestyle Program (PLP), which demonstrated effectiveness in improving weight, blood pressure, physical activity, and diet among NHPIs. The PPP consists of 8 lifestyle lessons and 4 SDOH activities delivered over a 3-month period.

The investigators will conduct an effectiveness-implementation hybrid type 2 trial using a 3 (Region) x 2 (Setting) x 2 (Delivery Mode) factorial design.

The long-term objective of this study is threefold:

1. To conduct an effectiveness-implementation hybrid 2 trial to test the effects of the PPP implementation strategies across different settings and modes of delivery among 600 NHPIs at risk for cardiometabolic-related conditions using an NHPI-approved and adapted evaluation framework. The investigators will also assess and compare the cost-effectiveness of the CHW-delivered PPP-Standard Facilitation and PPP-Enhanced Facilitation to support long-term sustainability.
2. To conduct a longitudinal Social Determinants of Health (SDOH) survey embedded within the trial to examine the reliability and validity of indices from 5 adapted SDOH instruments and to assess the associations between SDOH variables and chronic disease risk among NHPIs.
3. To implement and evaluate the contextually-based CHW training program on PPP delivery.

DETAILED DESCRIPTION:
Native Hawaiians and Pacific Islanders (NHPIs) continue to disproportionally experience high rates of cardiometabolic conditions, including obesity, hypertension, type 2 diabetes, and cardiovascular disease. To address these inequities, the Diabetes Prevention Program's Lifestyle Intervention (DPP-LI) was developed and subsequently culturally and contextually adapted into the PILI Lifestyle Program (PLP). Through consolidation and collaboration with NHPIs to revamp the DPP-LI, the original 16 lessons were modified into 8 lessons delivered over a 3-month period. These lessons offer empirically supported strategies, based on the Social Cognitive Theory, to improve healthy eating, physical activity, and time and stress management.

Community Health Workers (CHWs) serve as frontline public health workers and trusted community resources who can effectively disseminate and implement cardiometabolic-related interventions across diverse settings. The trusting relationship CHWs have with communities enables them to serve as a liaison and intermediaries between health, social, and cultural services and the community, facilitating access to services and improving their quality and cultural competence. NHPI CHWs are uniquely positioned to deliver effective interventions that improve cardiometabolic health outcomes and address their social determinants.

The PLP was adapted to include a Social Determinants of Health (SDOH) component and evaluated for its effectiveness in ClinicalTrials NCT06471595, resulting in what is now known as the PILI Pasifika Program (PPP).

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Native Hawaiian or Pacific Islander
* 18 years of age or older
* Have at least one of the following self-reported cardiometabolic conditions (Overweight or obesity defined as BMI ≥ 25, pre-diabetes or diabetes, high blood pressure, and/or high cholesterol)
* Able to do a moderate level of physical activity or exercise

Exclusion Criteria:

* Do not identify as Native Hawaiian or Pacific Islander
* Under 18 years of age
* Currently a student
* Do not have any of the following conditions (overweight/obesity, pre-diabetes/diabetes, high blood pressure, or high cholesterol)
* Have special dietary needs/dietary restrictions (due to cultural reasons and/or told by a healthcare provider)
* Pregnant women
* Have physical activity limitations/restrictions (told by a healthcare provider)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C | Assessment data will be collected at baseline, 3-month follow-up, and 9-month follow-up.
  A finger stick sample will be collected to measure hemoglobin A1C using the A1CNow+ kit.
Lipid Panel | Assessment data will be collected at baseline, 3-month follow-up, and 9-month follow-up.
  A fingerstick sample will be collected to measure Total Cholesterol, High-Density Lipoprotein (HDL), Low-Density Lipoprotein (LDL), and Triglycerides using the CardioChek Plus Analyzer.
Blood Pressure | Assessment data will be collected at baseline, 3-month follow-up, and 9-month follow-up.
  Systolic and diastolic blood pressure will both be measured by a digital blood pressure monitor device (Omron HEM-907XL IntelliSense).
Weight | Assessment data will be collected at baseline, 3-month follow-up, and 9-month follow-up.
  Weight will be calculated using a standardized mobile medical flat scale (Seca 876).

SECONDARY OUTCOMES:
Dietary Questionnaire | Assessment data will be collected at baseline, 3-month follow-up, and 9-month follow-up.
  A 5-item will be used to estimate the frequency and types of food a participant consumed in the past month. Taken directly from Common Survey IV, the dietary questionnaire consists of 5 items, documenting how many times per week in the past month participants have consumed specific types of food. The responses range from Never, 1-2 times per week, 3-4 times per week, 5-6 times per week, More than 6 times per week, and Don't know.
Brief Physical Activity Questionnaire | Assessment data will be collected at baseline, 3-month follow-up, and 9-month follow-up.
  A 2-item physical activity questionnaire will be used to briefly assess average physical activity behavior per week and the duration of the physical activity.
Food Literacy Form | Assessment data will be collected at baseline, 3-month follow-up, and 9-month follow-up.
  An 11-item questionnaire on food literacy will be used to ask participants' food literacy in regard to planning, managing, selecting, preparing, and eating healthy foods. The responses and scores range from 1-not at all/never, 2-disagree, 3-slightly disagree, 4-slightly agree, 5-yes/always. Higher scores indicate greater food literacy.
Social Connection and Isolation | Assessment data will be collected at baseline, 3-month follow-up, and 9-month follow-up.
  To assess how often social and emotional support is received. Responses range from Always, Usually, Sometimes, Rarely, and Never.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph K Kaholokula, PhD, Principal Investigator — University of Hawaii, Department of Native Hawaiian Health; Nia Aitaoto, PhD, Principal Investigator — National Association of Pasifika Organizations; Sheri-Ann Daniels, EdD, Principal Investigator — Papa Ola Lokahi
Locations (2):
- United States (2):
  - National Association of Pasifika Organizations, Fayetteville, Arkansas
  - Papa Ola Lokahi, Honolulu, Hawaii